CLINICAL TRIAL: NCT03218319
Title: Study of the Variations of the Blood Pressure After Nephrectomy for Renal Cancer
Brief Title: Study of the Variations of the Blood Pressure After Nephrectomy for Renal Cancer (VAPANCR)
Acronym: VAPANCR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 49RC17_0004
Record Dates: First submitted 2017-07-11; First posted 2017-07-14 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Renal Cancer; Nephrectomy; Blood Pressure
MeSH Terms: conditions — Kidney Neoplasms | interventions — Renin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental)
  Interventions: Biological: Renin measurement

INTERVENTIONS:
Biological: Renin measurement — patients will have a blood sample for measuring renin activity

SUMMARY:
This study evaluates the impact of nephrectomy in renal cancer on blood pressure and renal function. The patients will have a follow-up of their blood pressure and renal function until 6 months after their operation.

ELIGIBILITY:
Inclusion Criteria:

* Nephrectomy programmed for located renal cancer

Exclusion Criteria:

* Patients with metastatic renal cancer
* Incapacity to use a self-measurement tensiometer
* Patients treated for high blood pressure
* Patients with laxative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Blood pressure change | One time before the operation and twice after : 1 month and 6 months
  preoperative and postoperative measurements of blood pressure

SECONDARY OUTCOMES:
Renal function | One time before the operation and one after 6 months
  preoperative and postoperative measurements of renal function with measurements of renin activity and the glomerular filtration rate.
Cardiovascular risk | A clinical exam will perform before the surgery and 1 month and 6 months after
  Study the occurence of cardiovascular risk after nephrectomy